CLINICAL TRIAL: NCT03762161
Title: A Phase II Study of TAS-102 in Metastatic Platinum and Checkpoint Inhibitor-resistant Bladder Cancer
Brief Title: A Phase II Study of Lonsurf (TAS-102) in Metastatic Platinum and Checkpoint Inhibitor-resistant Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rahul Parikh (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Rahul Parikh, Principal Investigor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-TAS-102
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention TAS-102 (Experimental)
  Interventions: Drug: TAS 102

INTERVENTIONS:
Drug: TAS 102 — Participant self-administered orally at 35 milligrams per meter squared (mg/m2) twice daily Days 1-5 and 8-12 of every 28 day cycle

SUMMARY:
This study evaluates the clinical benefit of TAS-102 in participants with metastatic urothelial carcinoma who are resistant to cisplatin or carboplatin front-line and checkpoint inhibitors as second line therapy. All participants will receive TAS-102 in oral form twice per day on Days 1-5 and Days 8-12 of each 28 day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand this study, and participant willingness to sign a written informed consent.
* Participants must have histologically or cytologically confirmed locally advanced unresectable or metastatic urinary bladder (urothelial) cancer. Participants with mixed histologies are permitted as long as transitional cell carcinoma is present in the pathological specimen.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension
* Documented progression on or within 12 months of treatment with one previous platinum-containing regimen or ineligible to receive platinum-containing regimen. Neo-adjuvant or adjuvant platinum-based chemotherapy will be deemed to be first-line when participants progressed within 12 months of the last dose
* Documented progression on prior checkpoint inhibitor or ineligible to receive check-point inhibitor
* Adequate performance status, organ, and marrow function.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use two forms of adequate contraception.
* Men of child-bearing potential must not father a child or donate sperm while on this study and for 6 months after their last study treatment

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks of enrollment/registration.
* Current or anticipated use of other investigational agents while participating in this study.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding (if applicable).
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS 102.
* Patients with HIV on anti-retro-viral therapy with thymidine kinase substrates, for example, stavudine, zidovudine, telbivudine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia. Undergoing active treatment for a co-existing malignancy with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, thyroid cancer or incidental prostate adenocarcinoma detected at radical cystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (complete response+ partial response+ stable disease) | Up to 6 months
  Evaluated per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Progression-free survival rate (PFS) among participants | Up to 6 months
  Evaluated per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
Overall response rate (ORR) among participants | Up to 12 months
  Evaluated per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
Overall survival rate (OS) among participants | Up to 12 months
  Evaluated per Medical Record
Overall change in patient-reported quality of life outcomes | Up to 26 months
  Evaluated per Functional Assessment of Cancer Therapy - Bladder (FACT-Bl) version 4 - quality of life (QOL) questionnaire scores
  * FACT-Bl total score range is 0-156, derived by the sum of the sub-scales. Higher scores indicate better QOL.
  * FACT-Bl includes five sub-scales:
    * Physical Well-being (PWB), score range of 0-28
    * Social/Family Well-being (SWB), score range of 0-28
    * Emotional Well-being (EWB), score range of 0-24
    * Functional Well-being (FWB), score range of 0-28
    * Bladder Cancer Subscale (BlCS), score range of 0-48
  * Note: Negatively stated items are reversed by subtracting the response from "4".
Proportion of participants with Grade 3 or higher Adverse and Serious Adverse Events | Up to 26 months
  Evaluated per Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Parikh, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (2):
- United States (2):
  - University of Kansas Cancer Center - Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: Undecided